CLINICAL TRIAL: NCT03985579
Title: Influence of Kinesiology Taping Application on Severity of Signs and Symptoms in Breast Engorgement at Early Lactation Stage.
Brief Title: Influence of Kinesiology Taping Application on Severity of Signs and Symptoms in Breast Engorgement.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Żelazna Medical Centre, LLC (Other)
Responsible Party: Principal Investigator, Anna Jakóbik, Physiotherapist, Żelazna Medical Centre, LLC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 24/2019
Record Dates: First submitted 2019-06-05; First posted 2019-06-13 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Lactation Disorders
MeSH Terms: conditions — Lactation Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care and Kinesiology taping Group (Experimental): Application of elastic cotton strip with an acrylic adhesive that is used with the intent of treating pain and disability from athletic injuries and a variety of other physical disorders.
  Interventions: Other: Kinesiology taping application
- Standard care Group (No Intervention): Assistance in baby feeding, manual of device-assisted (lactator) milk expression, cold compress, ibuprofen, gentle breast massage, breathing and shoulder girdle exercise.

INTERVENTIONS:
Other: Kinesiology taping application — Application of elastic cotton strip with an acrylic adhesive that is used with the intent of treating pain and disability from athletic injuries and a variety of other physical disorders
  Arms: Standard care and Kinesiology taping Group

SUMMARY:
The aim of the research is to asses the efficacy of kinesiology taping application in breast engorgement in early postpartum stage.

Kinesiology application will be performed by women's health physiotherapist. Patient's perceived improvement and milk outflow following application will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* cesarian section or vaginal delivery
* delivery between 37 and 41 gestational week
* signs and symptoms of breast engorgement (significant increase of breast between 2nd and 10th day postpartum, pain, obstructed milk outflow)
* VAS 4 and more
* volume of milk outflow less than 20ml
* 6 point self-rated engorgement scale between 3 and 6

Exclusion Criteria:

* age less than 18 and more than 45
* patients after extensive surgical breast intervention or having breast implants
* allergy to kinesiology taping

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) change from baseline till 24 hours after intervention | assessment at the baseline 24 hours after intervention
  Pain assesment by Visual Analogue Scale (VAS scale), range 0-10, higher numbers represents worse outcome.
Human milk outflow change from baseline till 24 hours after intervention | assessment at the baseline and 24 hours after intervention
  Assesment of milk outflow based on infant body mass increase
6 point self-rated breast engorgement scale | assessment at the baseline
  assesment of breast engorgement, range 1-6, higher values represent worse outcomes
5 point perceived improvement scale | assessment 24 hours after intervention
  assessment of improvement of signs and symptoms of breast engorgement range 1-5, higher values represent worse outcomes
The Breastfeeding Self-Efficacy Scale | assessment at the baseline
  assessment of mother's attitude to breastfeeding

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) change from baseline till 3 hours after intervention | assessment at the baseline 3 hours after intervention
  Pain assesment by Visual Analogue Scale (VAS scale), range from 0-10, higher numbers represents worse outcome.
Human milk outflow change from baseline till 3 hours after intervention | assessment at the baseline and 3 hours after intervention
  Assesment of milk outflow based on infant body mass increase
5 point perceived improvement scale | assessment 3 hours after intervention
  assessment of improvement of signs and symptoms of breast engorgement, range 1-5, higher values represent worse outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Dorota Sys, PhD, Study Chair — Centre of Postgraduate Medical Education
Locations (1):
- Żelazna Medical Centre, St. Sophia Hospital, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zakarija-Grkovic I, Stewart F. Treatments for breast engorgement during lactation. Cochrane Database Syst Rev. 2020 Sep 18;9(9):CD006946. doi: 10.1002/14651858.CD006946.pub4. PMID 32944940